CLINICAL TRIAL: NCT01375166
Title: Coupling of Neural Activity and Retinal Blood Flow in Diabetes
Status: Terminated | Type: Observational
Why Stopped: not enough subjects recruited
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv. - Doz. Dr, Medical University of Vienna
Other Study IDs: OPHT-070111
Record Dates: First submitted 2011-04-11; First posted 2011-06-17 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diabetic retinopathy: Patients with early insulin dependent diabetes and no or mild non-proliferative retinopathy
- healthy: healthy control subjects

SUMMARY:
The prevalence of diabetes is increasing and the management of the disease is nowadays considered a major challenge. Affected patients have increased mortality and morbidity as well as a significant drop in the quality of life. The complications of diabetes can be classified as microvascular (e.g. nephropathy, neuropathy or retinopathy) or macrovascular (e.g. cardiovascular or cerebrovascular).

Several large-scale epidemiologic studies indicating that wider retinal venous caliber is strongly associated with the fasting glucose level as well as with diabetes. Another retinal vascular abnormality that is associated with diabetes is an abnormal retinal vascular response to flicker stimulation. Retinal vessel dilatation in response to stimulation with diffuse flicker light occurs due to a phenomenon called neurovascular coupling. This means that increased activity of neurons is associated with an increased retinal metabolism. This leads to a release of endogenous vasodilator substances and increased blood flow. However, previous studies were limited by the fact that retinal vessel diameters and blood flow were not measured simultaneously.

The present study aims to investigate whether the response of retinal vessel diameters and blood flow velocities to flicker stimulation is altered in patients with diabetes. Both parameters will be measured in real time using Fourier Domain Doppler OCT.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years, nonsmokers
* Normal findings in the medical history (except diabetes) and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* normal laboratory findings (except diabetes associated parameters) unless the investigator considers the abnormality to be clinically irrelevant
* normal ophthalmic findings (except mild diabetic retinopathy), Ametropia less than 6 diopters
* inclusion criterion of patients is type I diabetes with non or mild non-proliferative retinopathy

Exclusion criteria

Any of the following will exclude a healthy subject from the study:

* Regular use of vasoactive drugs
* Abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks
* History or presence of any ocular pathology
* History or family history of epilepsy
* Systemic hypertension defined as systolic blood pressure >150mmHg, diastolic blood pressure >90mmHg
* Pregnancy

Any of the following will exclude a subject with diabetes from the study:

* Presence of non-insulin dependent diabetes, maturity onset diabetes of the young (MODY diabetes)
* History or presence of any other diabetes induced vascular pathologies or any other ocular condition other then diabetic retinopathy
* Best corrected visual acuity <0.8
* Previous laser photocoagulation treatment
* Systemic hypertension defined as systolic blood pressure >150mmHg, diastolic blood pressure >90mmHg
* History or family history of epilepsy
* Abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 24 patients with early insulin dependent diabetes and no or mild non-proliferative retinopathy, non-smokers 24 age and sex matched healthy controls, non-smokers
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-03-06 (Actual); Primary Completion 2013-03-06 (Actual); Study Completion 2013-03-06 (Actual)

PRIMARY OUTCOMES:
Retinal vessel diameters | 18 months
Retinal blood flow velocities | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhöfer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria